CLINICAL TRIAL: NCT01484301
Title: The Impact of Opioid Tolerability Outcomes on the Management of Chronic Pain
Brief Title: Impact of Tolerability Issues on Chronic Pain
Status: Completed | Type: Observational
Sponsor: Janssen-Ortho Inc., Canada (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100408; NOCOMPOUNDNAP4001 (Other: Janssen-Ortho, Canada)
Record Dates: First submitted 2011-12-01; First posted 2011-12-02 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Pain
Keywords: Chronic pain; Opioids; Tolerability
MeSH Terms: conditions — Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study was to assess the impact of opioid tolerability-related issues experienced by Canadian chronic pain patients. Approximately 170 patients were enrolled from 16 recruiting centers across Canada. Eligible patients had a diagnosis of non-malignant, chronic pain requiring continuous use of strong opioids (>=4 days per week). Recruitment was initiated by physicians during routine care appointments at family or pain medicine practices. Patients were then directed to a website where they provided consent and completed an anonymized, password-protected, web-based survey that could be completed at home. This weekly online questionnaire was designed to document their chronic pain experience over a 12-week period. At the end of the 12-week study, physicians were asked to retrospectively complete information about pain treatments, over-the-counter (OTC) medication use for pain and opioid-related gastrointestinal (GI) side effects, as well as co-morbid conditions for each patient.

DETAILED DESCRIPTION:
This was a multi-center, non-interventional, observational study of patients receiving opioid treatment for chronic pain. Relevant Canadian data such as pain severity, treatment adherence, medical resource utilization, and interference with activities of daily living were collected to evaluate the impact of opioid-related side effects in chronic pain. The focus was mainly on side effects of the gastro-intestinal (GI) system. The study was divided into 2 components: a prospective, web-based patient survey and a physician-completed, retrospective chart review at study end. The patient survey included one baseline and 12 weekly follow-up surveys. The purpose of the web survey was to collect accurate data from the patient, particularly for outcomes that are not typically recorded in the medical charts, such as weekly pain severity scores, treatment adherence, and patient-reported outcomes (PROs), like medical resource use and impact on activities of daily living. To capture treatment management decisions, a retrospective chart review was performed by the physician or designee at the end of the 12-week period for each patient who completed baseline and at least one follow-up survey. Data collected included prescribed opioid and non-opioid medications for pain control, GI side effect treatments, co-morbid conditions/medications, and medical history. Eligible patients were offered an invitation letter at their usual care visit, where the study website was provided via weblink. Patients were nominally reimbursed for completing the survey. This study was reviewed and approved by an independent Ethics Committee, and informed consent was obtained from all patients. There was no study treatment, since this was a non-interventional, observational study that did not evaluate any J&J product; the duration of the study was 12 weeks of observation.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain of non-malignant origin (nociceptive, neuropathic or mixed pain types)
* Opioid requirement >=4 days per week, including new to opioids (<3 months exposure), opioid experienced (>3 months exposure), non-opioids or weak opioids (e.g., NSAIDS or Tramacet) for breakthrough or adjunctive use only
* Internet access; read/understand English or French.

Exclusion Criteria:

- Current or previous history of opioid addiction, abuse, or diversion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Family physician and pain medicine specialist practices
Sampling Method: Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2010-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Ortho, Canada Clinical Trial, Study Director — Janssen-Ortho Inc., Canada